CLINICAL TRIAL: NCT06979635
Title: Assessing the Safety, Performance, and User Experience of the Tandem Mobi Automated Insulin Delivery System Among Young Competitive Athletes in Real-world Settings.
Acronym: Captain MOBI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0800-24-RMC
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Competitive athletes; Hybrid Closed Loop System
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Tandem Mobi Hybrid Closed Loop (HCL) pump (Experimental): Tandem Mobi Hybrid Closed Loop (HCL) pump with an integrated Control-IQ algorithm (CIQ), the Dexcom G7 continuous glucose monitoring sensor (CGM ) and Tandem Mobi Mobile App
  Interventions: Device: Tandem Mobi Hybrid Closed Loop (HCL) pump

INTERVENTIONS:
Device: Tandem Mobi Hybrid Closed Loop (HCL) pump — Tandem Mobi Hybrid Closed Loop (HCL) pump with an integrated Control-IQ algorithm (CIQ), the Dexcom G7 continuous glucose monitoring sensor (CGM ) and Tandem Mobi Mobile App

SUMMARY:
A single arm, interventional study with 12 weeks study phase preceded by a 2-week run in phase, aiming to evaluate the effectiveness and applicability of the Tandem Mobi automated insulin delivery system (Tandem Mobi Pump System) for competitive youth athletes with type 1 diabetes in real-world conditions.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes (T1D) for at least 6 months
* 11≤Age≤18 years
* HbA1c <10.0%
* Current treatment with automated insulin delivery system (AID) or insulin pump for at least 1 month
* Willing to switch to Tandem Mobi Pump System and Dexcom CGM for the study duration
* Competitive-level athletes

Exclusion Criteria:

* Concomitant disease that influences metabolic control or HbA1c interpretation
* Individual has any unresolved adverse skin condition in the area of sensor or device placement (e.g., psoriasis, rash, Staphylococcus infection)
* Use of antidiabetic agents other than insulin
* Two or more episodes of severe hypoglycemia (hypoglycemia requiring treatment by another person) within the previous 6 months
* One or more episodes of ketoacidosis requiring hospitalization within 6 months prior to screening
* Individual has a positive pregnancy screening test

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Sensor glucose percentage of time in range (70-180 mg/dl) | At the end of the 12 weeks intervention period

SECONDARY OUTCOMES:
Percentage of sensor glucose readings <54 mg/dl | At the end of the 12 weeks intervention period
Percentage of sensor glucose readings >180 mg/dl | At the end of the 12 weeks intervention period
Percentage of sensor glucose readings >250 mg/dl | At the end of the 12 weeks intervention period
HbA1c | At the end of the 12 weeks intervention period

OTHER OUTCOMES:
Serious Adverse Events (SAE) | At the end of the 12 weeks intervention period
Diabetic Ketoacidosis (DKA) events | At the end of the 12 weeks intervention period
Severe Hypoglycemia events | At the end of the 12 weeks intervention period
Percentage of sensor glucose readings in the range 70 to 140 mg/dL | At the end of the 12 weeks intervention period
Percentage of sensor glucose readings in the range 70 to 180 mg/dL | At the end of the 12 weeks intervention period
Percentage of sensor glucose readings >180 mg/dL | At the end of the 12 weeks intervention period
CGM derived indices- Mean glucose | At the end of the 12 weeks intervention period
CGM derived indices: Coefficient of variation | At the end of the 12 weeks intervention period
CGM derived indices: Peak glucose and change in glucose from the start of the meal to the peak (only calculated for post-meal periods) | At the end of the 12 weeks intervention period
CGM derived indices: change in glucose from the start of the exercise to the nadir. | At the end of the 12 weeks intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Marie Muller, MD, Principal Investigator — Schneider Children's Medical Center
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel